CLINICAL TRIAL: NCT02125890
Title: The Effect of Tranexamic Acid in Ruptured Abdominal Aortic Aneurysms
Brief Title: Effect of Tranexamic Acid in Ruptured Abdominal Aortic Aneurysms
Acronym: TARAA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB-13-91
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Abdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tranexamic Acid (Experimental): We will be administering Tranexamic Acid in patients with ruptured abdominal aortic aneurysms to determine if this has an effect on primary outcome measures as significant bleeding, blood transfusion requirements.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — two doses of Tranexamic Acid will be given to patients with rupture abdominal aortic aneurysms
  Other Names: Cyklokapron

SUMMARY:
An abdominal aortic aneurysm occurs when the part of the aorta travelling down into the abdomen balloons out more than 50%. If caught early, treatments can be used to prevent rupture of the aneurysm. However, many of these aneurysms are asymptomatic and go undetected until they rupture, causing large amounts of blood to spill into the abdominal cavity and typically leads to death, if left untreated. The current mortality rate is between 50 and 90%. The resources required to treat patients with ruptured aortic aneurysms is quite substantial given that they need blood transfusions and can have prolonged hospital stays. Patients either undergo a more invasive operative repair, associated with greater blood products transfusions and complications, or if relatively stable, undergo a less invasive repair with tubes called stents. There is less morbidity associated with the latter, endovascular repair. To prevent blood loss in elective surgeries, drugs that promote blood clotting are often used. One drug, tranexamic acid , has been shown to reduce blood loss, reduce the number of blood transfusions required and improve patient outcomes in elective cardiac and orthopaedic surgeries, and more recently, in patients with traumatic hemorrhage. However, this drug has not been tested in this particular population. The purpose of this pilot project is to evaluate the effectiveness of tranexamic acid in reducing clinically significant bleeding in patients with ruptured aortic aneurysms in hospital sites across Saskatchewan using a single-group intervention design. The investigators will compare the data from patients treated with tranexamic acid to retrospective data from a control group that is matched on key variables. The investigators predict that tranexamic acid will result in reduced bleeding, reduced need for blood transfusions, less patients that require open surgery and improved patient outcomes. The results of this study will help determine if this treatment is effective at preventing the death of many people with ruptured abdominal aortic aneurysms.

DETAILED DESCRIPTION:
The primary purpose of this study is to examine the effectiveness of TXA in reducing clinically significant bleeding in a novel patient population (ruptured AAA). The first phase of this study will involve a small pilot project, consisting of ~25 patients who will be administered TXA during their treatment for a ruptured AAA. We will compare the amount of clinically significant bleeding from a group of patients treated prospectively with TXA to data collected retrospectively over the previous year from a matched control group of patients who were treated for a ruptured AAA but not given TXA. At the conclusion of this pilot, if the data reveal that administration of TXA in patients with ruptured AAA reduces the incidence of clinically significant bleeding, then we will proceed to a multicenter national trial to determine the generalizability of TXA use to treat ruptured AAA in patients across Canada.

METHODOLOGY This study employs a 1-year prospective non-randomized intervention design. All patients that present to a southern Saskatchewan hospital with a clinically-confirmed ruptured AAA during the 1-year enrollment period will be potential participants. We aim to enroll 25 consecutive patients with ruptured AAA.

Regina (Regina General Hospital) is the primary site for this study. Rural hospitals in the surrounding area that refer patients to Regina for trauma surgery will be the secondary sites. Local Health Canada Qualified Investigators will be responsible for the managing the study at each hospital

Diagnosis Patients presenting to a Saskatchewan emergency room (ER) with symptoms of a ruptured AAA might have an ultrasound or CT scan to confirm diagnosis as part of investigations. The current standard of care, however, is clinical assessment, which may be aided by prior imaging history of an unruptured AAA. Enrollment without radiologic confirmation at the time of presentation to the ER would take place upon the recommendation of the vascular surgeon in Regina. At that time, the patient's pharmaceutical history will be examined using the Pharmaceutical Information Program (PIP) system to determine if the patient has any contradictions to TXA as listed above for patients in Saskatchewan. Since other provinces do not have the PIP program, the study will be restricted to patients with Saskatchewan Health Cards.

For patients that meet the study inclusion criteria and none of the exclusion criteria, we will proceed with a three-part informed consent procedure based on the individual case (i.e., patient is conscious and capable of giving informed consent, patient is incapable of giving informed consent so the patient's next-of-kin or legally authorized representative will provide verbal or written consent, or patient is incapable of giving consent and there is no next-of-kin or legally authorized representative that can be contacted in a timely manner (30 minutes) so "Dual Physician Consent" will be used).

TXA Administration Patients who have an ultrasound or CT in a hospital/care centre outside of the catchment area Regina (rural patients) will receive the first dose of TXA (one gram IV over ten minutes) by the local attending physician (ER or family physician). For patients who are diagnosed in Regina, the vascular surgeon will be responsible for ordering TXA upon diagnosis in the emergency room. Rural patients in the Regina catchment area will then be transferred to the trauma center in Regina and the vascular surgeon will be notified that the patient is part of the study and has received TXA. For all patients, the second dose of TXA (one gram IV will be administered over 8 hours) will be ordered by the vascular surgeon or anesthesiologist in the ER, the OR theatre or the intensive care unit in Regina. Dosing recommendations are based on data resulting from the CRASH-2 Trial.30

If the patient stabilizes as a result of the TXA administration, the patient will proceed to the angiogram suite (interventional radiology) where a vascular surgeon will perform endovascular stenting. If the patient becomes or remains hemodynamically unstable after arrival, the patient will proceed to the operating room for laparotomy and open repair of the aneurysm. Procedures and subsequent treatment will remain the same as the current standard of care for ruptured AAA's. We will only collect data on the patient and his/her care during the patient's stay in hospital. Given that there is little risk of adverse events occurring from administration of TXA after hospital stay, once the patient has been released from hospital, there will be no direct follow-up.

Statistical analysis We will compare data from the experimental group (TXA) to the data from the matched control patients collected retrospectively (controls). The patients will be matched on age, sex, ethnicity, history of peripheral vascular disease, coronary artery disease, aneurysms, and current medications (antihypertensives, anticoagulants, NSAIDs). Our primary analyses will compare outcomes that are measured on interval/ratio scales using independent t-tests or ANOVA's or non-parametric Mann-Whitney/Kruskal-Wallis if the data are skewed. For categorical data, chi-square or Fisher's Exact tests with effect size measures will be used to analyze the relationship between treatment and outcome (e.g. incidence of abdominal compartment syndrome in experimental vs. control group). We will use two-sided tests with alpha set at .05 to be able to detect if TXA produces worse outcomes than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* any patient with a ruptured aortic aneurysm, regardless of sex, age, ethnicity who may or may not be on anticoagulant or anti-platelet medications for comorbid conditions.

Exclusion Criteria:

* pregnancy
* hypersensitivity to Tranexamic Acid (TXA)
* acquired defective colour vision
* active intravascular clotting or disseminated intravascular clotting (DIC)
* subarachnoid hemorrhage
* thromboembolic disease
* age < 18 years of age
* known clotting disorder
* patients receiving thrombin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-07; Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Clinically significant bleeding | Participants will be followed for average length of stay, which is approximately two weeks
  Hemoglobin less than 100 g/L or 2 or more units of red blood cells or 2 or more units of fresh frozen plasma (FFP), or 5 or more units of cryoprecipitate, or more than 1 unit of platelets, or activation of the health region's Massive Transfusion Protocol.

SECONDARY OUTCOMES:
Number of ruptured abdominal aortic aneurysms requiring open laparotomy compared to endovascular stunting | Patients will be followed during hospital length of stay, which is an average of two weeks
  We will compare the number of ruptured aortic aneurysms that require open repair with laparotomy versus those that can proceed with endovascular stenting.
Number of blood transfusions | Patients will be followed during hospital length of stay, an average of two weeks
  We will examine the number of blood transfusions, including individual products
Incidence of Transfusion Related Acute Lung Injury (TRALI) | Patients will be followed during hospital length of stay, which is an average of two weeks
  TRALI refers to acute lung injury associated with transfusion of blood and blood products
Incidence of Transfusion Related Reactions | Patients will be followed during hospital length of stay, which is an average of two weeks
  This will examine the incidence of transfusion related reaction in patients with ruptured aneurysms
Mechanical ventilator days | Patients will be followed during hospital length of stay, an average of two weeks
  The number of days required by the patient on a ventilator will also be examined.
Length of stay in ICU | Patients will be followed during hospital length of stay, an average of two weeks
  Determination of length of stay in ICU
Length of stay in hospital | Patients will be followed during hospital length of stay, an average of two weeks
  Determination of length of stay in hospital
Incidence of intrabdominal hypertension | Patients will be followed during hospital length of stay, an average of two weeks
  Incidence of intrabdominal hypertension may be related to blood products and resuscitation requirements.
Incidence of Abdominal Compartment Syndrome (ACS) | Patients will be followed during hospital length of stay, an average of two weeks
  We will examine the incidence of abdominal compartment syndrome (ACS)
Requirement of either continuous or intermittent renal replacement therapy (dialysis) | Patients will be followed during hospital length of stay, an average of two weeks
  If patients are hypotensive (low blood pressure), they will require vasoactive or inotropes for maintenance of blood pressure. These patients would not tolerate conventional intermittent hemodialysis. Instead, in this group, Continuous Renal Replacement Therapy would be the option. If the patient has normal blood pressure, and is not on vasoactive drugs, then intermittent renal replacement therapy would be acceptable.
Cardiac morbidity | Patients will be followed during hospital length of stay, an average of two weeks
  Cardiac morbidity such as cardiac arrest, myocardial infarction, stroke or seizure will be examined
Multiorgan Dysfunction Score | Patients will be followed during hospital length of stay, an average of two weeks
  A scoring system that measures dysfunction in six organ systems.
All cause 28 day mortality | 28 days post-surgery
  We will assess all cause 28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jagadish Rao, MD, FRCSC, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Jagadish Rao, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No